CLINICAL TRIAL: NCT04337983
Title: Hemodynamic Characteristics of Patients With SARS-CoV-2: PiCCOVID Study
Brief Title: Hemodynamic Characteristics of Patients With SARS-CoV-2
Acronym: PiCCOVID
Status: Completed | Type: Observational
Sponsor: Bicetre Hospital (Other)
Responsible Party: Principal Investigator, Xavier Monnet, Professor Xavier Monnet MD. PhD., Bicetre Hospital
Other Study IDs: 2020-A00793-36
Record Dates: First submitted 2020-03-30; First posted 2020-04-08 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Coronavirus; SARS-CoV-2; COVID-19; Acute Respiratory Distress Syndrome; Shock; Acute Circulatory Failure; Left Ventricular Dysfunction; Fluid Overload
Keywords: Hemodynamic chracteristics; Transpulmonary thermodilution; Preload-dependency; Echocardiography; Extravascular lung water; Pulmonary vascular permeability index
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Respiratory Distress Syndrome; Shock; Ventricular Dysfunction, Left; Edema | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Transpulmonary thermodilution — Obtained by averaging the results of three thermodilution measurements. Each thermodilution is performed by injecting a bolus (15 mL) of cold saline (less than 10°C)
Device: Echocardiography — Daily echocardiography evaluation

SUMMARY:
The outbreak of coronavirus disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has been declared a public health emergency of international concern. Hospitalized COVID-19-positive patients requiring ICU care is increasing along with the course of epidemic. A large number of these patients developed acute respiratory distress syndrome (ARDS) according to current data. However, the related hemodynamic characteristic has so far been rarely described.

DETAILED DESCRIPTION:
The outbreak of COVID-19 is a worldwide concern. To our knowledge, the details of the hemodynamic characteristics of COVID-19 patients have not yet been well described. Besides, the cardiac injury was reported in about 7-17% of hospitalized patients with COVID-19 in previous Chinese publications and is much more common in patients admitted to ICU and non-survivors. However, no systematic assessment, including echocardiography evaluating the left ventricular function of these patients has been declared. In addition, extravascular lung water (EVLW) and pulmonary capillary permeability are two hall markers in ARDS patient's management, and transpulmonary thermodilution is a validated method to provide these values at the bedside. However, no study has reported the characteristic profile of these variables during ARDS caused by SARS-Cov2. A better knowledge of these characteristics would also be helpful in guiding their management.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed or suspected SARS-Cov2 cases
* Patients admitted to ICU, defined as a unit in which patients can receive vasopressors.
* Monitored by a transpulmonary thermodilution system (PiCCO2 (Pulsion Medical Systems, Feldkirchen, Germany) or EV1000 (Edwards Lifesciences, Irvine, United States of America).

Exclusion Criteria:

* SARS Cov-2 Negative
* Refusal to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: SARS-Cov2 positive patients admitted to ICU and monitored by transpulmonary thermodilution system will be included.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Body temperature | Through study completion, an estimation of 6 months
  Body temperature(°C)
Blood pressure | Through study completion, an estimation of 6 months
  Blood pressure in mmHg
Pulse (heart rate) | Through study completion, an estimation of 6 months
  Pulse (heart rate) in times/minute
Respiratory rate | Through study completion, an estimation of 6 months
  Respiratory rate in times/minute
Data provided by transpulmonary thermodilution-CI | Through study completion, an estimation of 6 months
  Cardiac index (L/min/m2)
Data provided by transpulmonary thermodilution-GEDV | Through study completion, an estimation of 6 months
  Global end-diastolic volume(mL/m2)
Data provided by transpulmonary thermodilution-EVLW | Through study completion, an estimation of 6 months
  Extravascular lung water (mL/kg)
Data provided by transpulmonary thermodilution-PVPI | Through study completion, an estimation of 6 months
  Pulmonary vascular permeability index
Incidence of abnormal laboratory test results | Through study completion, an estimation of 6 months

SECONDARY OUTCOMES:
Incidence of new-onset or reversible systolic left ventricular dysfunction | Through study completion, an estimation of 6 months
  Left ventricle ejection fraction, Segmental left ventricle contractility, Speckle tracking data of the left and right ventricles, Dimensions of right and left cavities and Diastolic function of left ventricle
Changes of extravascular lung water measured by transpulmonary thermodilution | Change from baseline extravascular lung water at 6 months
  The worst extravascular lung water
Changes of pulmonary vascular permeability index measured by transpulmonary thermodilution | Change from baseline extravascular lung water at 6 months
  The worst pulmonary vascular permeability index
Correlation between the hemodynamic characteristics and 90-day mortality | Up to 90th day after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Bicetre Hospital, Paris, Val-de-Marne, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Driggin E, Madhavan MV, Bikdeli B, Chuich T, Laracy J, Biondi-Zoccai G, Brown TS, Der Nigoghossian C, Zidar DA, Haythe J, Brodie D, Beckman JA, Kirtane AJ, Stone GW, Krumholz HM, Parikh SA. Cardiovascular Considerations for Patients, Health Care Workers, and Health Systems During the COVID-19 Pandemic. J Am Coll Cardiol. 2020 May 12;75(18):2352-2371. doi: 10.1016/j.jacc.2020.03.031. Epub 2020 Mar 19. PMID 32201335
- [Background] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Schuster DP. The search for "objective" criteria of ARDS. Intensive Care Med. 2007 Mar;33(3):400-2. doi: 10.1007/s00134-006-0499-5. Epub 2007 Jan 13. No abstract available. PMID 17221188
- [Background] Jozwiak M, Silva S, Persichini R, Anguel N, Osman D, Richard C, Teboul JL, Monnet X. Extravascular lung water is an independent prognostic factor in patients with acute respiratory distress syndrome. Crit Care Med. 2013 Feb;41(2):472-80. doi: 10.1097/CCM.0b013e31826ab377. PMID 23263578
- [Background] Monnet X, Teboul JL. Transpulmonary thermodilution: advantages and limits. Crit Care. 2017 Jun 19;21(1):147. doi: 10.1186/s13054-017-1739-5. PMID 28625165
- [Derived] Shi R, Lai C, Teboul JL, Dres M, Moretto F, De Vita N, Pham T, Bonny V, Mayaux J, Vaschetto R, Beurton A, Monnet X. COVID-19 ARDS is characterized by higher extravascular lung water than non-COVID-19 ARDS: the PiCCOVID study. Crit Care. 2021 Jun 1;25(1):186. doi: 10.1186/s13054-021-03594-6. PMID 34074313